CLINICAL TRIAL: NCT05758493
Title: Characterizing Iodine-124 Evuzumitide (AT-01) in Systemic Amyloidosis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Attralus, Inc. (Industry)
Responsible Party: Principal Investigator, Ahmad Masri, Associate Professor, Oregon Health and Science University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 24299
Record Dates: First submitted 2023-01-25; First posted 2023-03-07 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Amyloidosis; Transthyretin Amyloidosis
MeSH Terms: conditions — Amyloidosis; Amyloidosis, Hereditary, Transthyretin-Related

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients with ATTR-CM (Experimental): Patients with ATTR-CM will undergo hybrid 124I-Evuzamitide PET/MRI imaging (or PET/CT) at baseline and in a subgroup, repeat imaging will be performed at an interval of 6-12 months.
  Interventions: Diagnostic Test: 124I-Evuzamitide

INTERVENTIONS:
Diagnostic Test: 124I-Evuzamitide — Amyloid reactive protein used as imaging agent to detect systemic amyloidosis
  Other Names: AT-01

SUMMARY:
This is a single center prospective study evaluating 124I-evuzumitide in patients with systemic amyloidosis. The purpose of this study is to 1)identify and characterize the distribution and uptake of 124I-evuzumitide in patients with transthyretin amyloid cardiomyopathy (ATTR-CM) and 2) Correlate the uptake with the structure and function of different organs, including the heart. To achieve these goals, eligible patients will undergo primarily hybrid positron emission tomography and magnetic resonance imaging (PET/MRI). In a subgroup of patients who are unable to undergo PET/MR, computed tomography will be used instead of MRI (i.e. PET/CT). In a subgroup of patients, repeat imaging with the same modality will be done at a interval of 6-12 months. Clinically available data (demographics, phenotype, imaging, laboratory) will also be collected to characterize the disease in each patient.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will at least have one of the following conditions: systemic amyloidosis with known organ involvement, carrier of a known pathogenic mutation in the transthyretin gene, multiple myeloma, and monoclonal gammopathy of undetermined significance
2. Patient willing to consent for the study and undergo the study procedures.

Exclusion Criteria:

1. Has severe claustrophobia or any medical condition that would prevent completion of the imaging protocol
2. Has a known allergy to potassium iodide treatment or to gadolinium.
3. Patients on dialysis or those with eGFR <30 cc/min/1.73 m2 will be excluded from undergoing gadolinium-enhanced cardiac MRI.
4. Has received heparin or heparin analogs (e.g., enoxaparin, dalteparin, fondaparinux) within 7 days prior to 124I-Evuzumitide administration

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-01-10 (Actual); Primary Completion 2027-12-10 (Estimated); Study Completion 2028-03-10 (Estimated)

PRIMARY OUTCOMES:
Correlation between ECV and 124I-Evuzamitide cardiac uptake and distribution | At baseline scan
  Pearson Correlation Coefficient of ECV (%) and SUV (124I-Evuzamitide) globally and at a per segment basis

SECONDARY OUTCOMES:
Correlation between clinical cardiac biomarkers (i.e. stage of amyloidosis) and myocardial 124I-Evuzamitide uptake | At baseline scan
  Pearson Correlation Coefficient of stage of amyloidosis (Mayo Staging System) and SUV (124I-Evuzamitide)
Correlation between Kansas City Cardiomyopathy Questionnaire overall summary score (KCCQ-OS) and myocardial 124I-Evuzamitide | During baseline scan and follow up scan
Correlation between New York Heart Association (NYHA) class and 124I-Evuzamitide uptake | During baseline scan and follow up scan
Correlation between liver and spleen ECV and their respective 124I-Evuzamitide uptake | During baseline scan and follow up scan
Proportion of patients with ATTR-CM and MGUS or smoldering myeloma who are correctly classified as ATTR-CM based on 124I-Evuzamitide distribution and uptake | During baseline scan

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wall JS, Martin EB, Endsley A, Stuckey AC, Williams AD, Powell D, Whittle B, Hall S, Lambeth TR, Julian RR, Stabin M, Lands RH, Kennel SJ. First in Human Evaluation and Dosimetry Calculations for Peptide 124I-p5+14-a Novel Radiotracer for the Detection of Systemic Amyloidosis Using PET/CT Imaging. Mol Imaging Biol. 2022 Jun;24(3):479-488. doi: 10.1007/s11307-021-01681-2. Epub 2021 Nov 16. PMID 34786667